CLINICAL TRIAL: NCT00423280
Title: A Randomised, Placebo-Controlled Study of Two Doses of Oral 6R-BH4 on Vascular Function in Subjects With Coronary Artery Disease
Brief Title: Effect of 6R-BH4 Treatment in Coronary Artery Disease (OXBIO Study)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Mrs Heather House, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06/Q1604/114
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease
Keywords: Endothelium; Nitric Oxide; Magnetic Resonance Imaging; Tetrahydrobiopterin
MeSH Terms: conditions — Coronary Artery Disease | interventions — sapropterin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 700mg/day 6R-BH4
  Interventions: Drug: 6R-BH4
- 2 (Active Comparator): 400mg/day 6R-BH4
  Interventions: Drug: 6R-BH4
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: 6R-BH4

INTERVENTIONS:
Drug: 6R-BH4 — 6R-BH4 tablets 700mg/day, 6R-BH4 tablets 400mg/day or placebo
  Other Names: Sapropterin dihydrochloride

SUMMARY:
The purpose of this study is to determine the effect of 6R-BH4 on vascular function in patients with coronary artery disease. We hypothesize that 6R-BH4 will improve vascular function in these patients.

DETAILED DESCRIPTION:
Decreased production of nitric oxide (NO) from the endothelium (the layer of cells that forms the lining of all blood vessels) has been shown to contribute to atherosclerosis. NO has multiple beneficial effects on vascular function. Endothelial function can be measured in humans via a number of methods, and endothelial dysfunction has been shown to be a strong adverse predictor of cardiovascular events and mortality.

Tetrahydrobiopterin (BH4) is essential for the production of NO in endothelial cells. 6R-BH4 is a synthetic version of naturally occurring BH4. We aim to investigate the effects of oral 6R-BH4 supplementation on endothelial function in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Multi-vessel coronary artery disease scheduled for coronary artery bypass surgery (CABG)

Exclusion Criteria:

* Inability to provide informed consent
* Female subject who is pregnant, lactating or planning pregnancy during course of study
* Prior clinical diagnosis of heart failure requiring diuretic therapy with evidence of severe left ventricular dysfunction
* Recent acute coronary event (<4 weeks)
* Emergency CABG
* Newly diagnosed diabetes mellitus (<1 month)
* Body weight >130kg
* Impaired renal function (creatinine >180umol/l)
* Elevated liver function tests (ALT >50umol/l or AST >2x normal)
* Pacemakers, ICDs or metallic implants not compatible with MRI scanning
* Subjects receiving experimental medications or participating in another study
* Terminally ill subjects
* Known hypersensitivity to 6R-BH4
* Concomitant treatment with methotrexate, levodopa, PDE-3 or PDE-5 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Vascular function using non-invasive magnetic resonance imaging (MRI). | Pre- and post- treatment with 6R-BH4 or placebo

SECONDARY OUTCOMES:
Laboratory measures of vascular function. | At time of CABG surgery

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Channon, MD FRCP, Principal Investigator — University of Oxford
Locations (1):
- Department of Cardiovascular Medicine, University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Cunnington C, Van Assche T, Shirodaria C, Kylintireas I, Lindsay AC, Lee JM, Antoniades C, Margaritis M, Lee R, Cerrato R, Crabtree MJ, Francis JM, Sayeed R, Ratnatunga C, Pillai R, Choudhury RP, Neubauer S, Channon KM. Systemic and vascular oxidation limits the efficacy of oral tetrahydrobiopterin treatment in patients with coronary artery disease. Circulation. 2012 Mar 20;125(11):1356-66. doi: 10.1161/CIRCULATIONAHA.111.038919. Epub 2012 Feb 7. PMID 22315282
- [Derived] Cunnington C, Channon KM. Tetrahydrobiopterin: pleiotropic roles in cardiovascular pathophysiology. Heart. 2010 Dec;96(23):1872-7. doi: 10.1136/hrt.2009.180430. Epub 2010 Sep 13. PMID 20837663